CLINICAL TRIAL: NCT05927077
Title: EXPOSO-METER - Characterizing the Environmental and Human Exposome of Mixtures of Pollutants at High Trophic Levels
Brief Title: Chemometers to Determine the Environmental and Human Exposome by Mixtures of Pollutants
Acronym: EXPOSO-METER
Status: Not yet recruiting | Type: Observational
Sponsor: Helmholtz Centre for Environmental Research - UFZ (Other)
Collaborators: Duke University (Other); Seoul National University (Other); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: EXPOSO-METER
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Exposure to Pollution

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Lipid tissue and blood of the study participants will be collected, in which the investigators will determine patterns of chemicals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy study participants who undergo planned surgeries for weight reduction from Central Europe: The investigators will take benefit of planned surgeries for weight reduction to collect study material that allows to determine the chemical exposome of the participants
  Interventions: Procedure: planned surgery for weight reduction
- healthy study participants who undergo planned surgeries for weight reduction from North America: The investigators will take benefit of planned surgeries for weight reduction to collect study material that allows to determine the chemical exposome of the participants
  Interventions: Procedure: planned surgery for weight reduction
- healthy study participants who undergo planned surgeries for weight reduction from South Korea: The investigators will take benefit of planned surgeries for weight reduction to collect study material that allows to determine the chemical exposome of the participants
  Interventions: Procedure: planned surgery for weight reduction

INTERVENTIONS:
Procedure: planned surgery for weight reduction — planned surgeries will be used to collect study material to determine chemical patterns in the study participants from the different geographical regions

SUMMARY:
Motivation of this study

Human life is full of chemicals: They support the provision of cure, clothes, shelter, transportation and even nourishment of the world population. But can they also represent a risk for humans? Many of these chemicals can be taken up into the human body. Often, they are transformed and excreted directly, but some chemicals persist over longer time periods or accumulate in living organisms. Since there are many thousands of chemicals in the environment and products humans use on a daily basis, there may be complex mixtures around, and consequently also in the human body. The investigators start a new project at the Helmholtz Centre for Environmental Research (UFZ) in Leipzig, Germany. It is called EXPOSO-METER and attempts to make these chemicals measurable in an easy and comparable way, to better characterize this potential hazard. With the valuable contribution of the participants and collaborators, the investigators will be able to describe and compare the situation for similar groups of study participants in Central Europe, North America and Asia. The aim is to characterize the chemicals and see which potential effects their presence may have. In the project, the investigators will also compare human samples to material from the environment, e.g., seal and fox samples, to improve the understanding of the occurrence and fate of chemicals in the environment and in the human body.

DETAILED DESCRIPTION:
Determination of sample size

The research project EXPOSO-METER does not aim for a large cohort study but for a proof-of-concept pilot study that will form the basis for future work. Therefore, two approaches were followed to determine the sample size:

1. Based on a literature review of similar studies, a closely matching example from a high-level journal was identified. It worked with 16 individuals in total from two German cities (different tissues, in total 88 samples). The work in EXPOSO-METER will by far exceed this number of study participants. Furthermore, three global regions are expected to show explicit large-scale differences due to distinct lifestyle and exposure conditions in the U.S., Europe and South Korea.
2. Cochran's formula [n= (Z^2 p(1-p))/e^2] was applied for sample size calculation: with a 90 percent confidence level (Z=1.645), maximum variability (50 percent, i.e., p=0.5) and +/-10 percent precision (e=0.1), it renders a minimum sample size of 68 participants.

As a combined result, the minimum sample size is therefore 50 study participants per region, with 100 study participants being ideal per region.

Sample collection

The following distribution of study participants is targeted: 25 female and 25 male participants of 30-40 years, and 5 female and 5 male participants of each of these age groups: 20-30, 40-50, 50-60, 60-70, 70-80 years. The following samples are collected: (1) 2-20 g of excized subcutaneous lipid from the lower abdomen, placed in a glass vial labelled with a unique sample identification number (ID) and stored at -20 °C; (2) 5 mL of blood using a tube filled with the complexation agent ethylenediaminetetraacetic acid (EDTA) and labelled with the ID and stored at -20 °C. In addition, the study participants are asked to fill the participants' questionnaire to be labelled with the ID. Once complete, the sample set is shipped to the UFZ laboratories.

Sample processing at UFZ

Lipid tissue: Samples will be thawed, homogenized and its lipid content determined. (a) Passive equilibrium sampling: To the sample, silicone thin-film samplers are added, which are medical grade silicone sheets of a suitable size and thickness, precleaned using Soxhlet extraction with ethyl acetate. After approx. 48 h (required for equilibration) the silicone is removed, its surface cleaned thoroughly and the chemicals from the silicone are extracted with ethyl acetate. (b) Total extraction: A subsample of the lipid tissue will be extracted directly with different mixtures of solvents. The solvent from both approaches is evaporated, the samples are cleaned via a range of columns, and the chemicals are analyzed by gas/liquid chromatography (GC/LC) coupled to high-resolution mass spectrometry (HRMS) or tandem mass spectrometry (MS/MS). In total, 150 + 400 chemicals will be screened for using the two techniques. For quality assurance/quality control, stable isotope-labelled internal standard compounds are used. The results will be set into context across regions, and data from the questionnaires will be used to support data interpretation.

Blood: The blood samples will be submitted to an extraction procedure currently under development, similar to the approaches described above, the extracts are cleaned, concentrated and analyzed by GC/LC-HRMS (or MS/MS), as described above.

Possible extensions

As a first option to further extend this work, the investigators aim to explore non-targeted screening of the broad mixtures of chemicals that are quantified in a targeted mode at UFZ. Likely there are many more chemicals, yet unidentified, that would be of interest to study, either at UFZ, via the EXPOSO-METER collaboration or via other related projects. For other projects, written consent will be sought before starting the work.

As a second option, the investigators would be interested in adding to the chemical profiling described above by exploring the application of bioanalytical tools (bioassays) to characterize the mixture effects elicited by the complex array of chemicals present in the human samples. This could either be done at UFZ, via the EXPOSO-METER collaboration or via other future projects. For other projects, written consent will be sought before starting the work.

ELIGIBILITY:
Inclusion Criteria:

* willingness to contribute to the EXPOSO-METER research
* cover geographical patterns
* cover all sexes and age groups to derive patterns

Exclusion Criteria:

* none

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The core group undergoing surgeries for weight reduction are between 30 and 40 years old. Hence, the following distribution of study participants is targeted: 25 female and 25 male participants of 30-40 years, and 5 female and 5 male participants of each of these age groups: 20-30, 40-50, 50-60, 60-70, 70-80 years.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Patterns of the human exposome in three global regions | samples will be collected only on the very same day when the planned surgery is carried out, questionnaires will be filled in the same context
  A wide range of chemicals will be determined in the human tissue and blood samples. In total, 150 + 400 chemicals are analyzed by gas/liquid chromatography (GC/LC) coupled to high-resolution mass spectrometry (HRMS) or tandem mass spectrometry (MS/MS) following the sample treatment described above. The resulting data will be used to describe and compare the patterns across geographical scales, and correlations of the observed chemical patterns with different characteristics of the study participants (such as age, sex, height, weight, and certain lifestyle factors (e.g. smoking status, nutritional aspects) etc.) will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Helmholtz-Centre for Environmental Research - UFZ, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
We plan to fully anonymize the data, details are checked by the data protection officers (DPOs) of the participating institutions. Only information on age, sex, height, weight, and certain lifestyle factors (e.g. smoking status, nutritional aspects) will be used for data interpretation.

REFERENCES:
- [Background] Baumer A, Jasch S, Ulrich N, Bechmann I, Landmann J, Stover A, Escher BI. Chemical mixtures in human post-mortem tissues assessed by a combination of chemical analysis and in vitro bioassays after extraction with silicone. Environ Int. 2021 Dec;157:106867. doi: 10.1016/j.envint.2021.106867. Epub 2021 Sep 16. PMID 34537519
- [Result] Reiter EB, Escher BI, Siebert U, Jahnke A. Activation of the xenobiotic metabolism and oxidative stress response by mixtures of organic pollutants extracted with in-tissue passive sampling from liver, kidney, brain and blubber of marine mammals. Environ Int. 2022 Jul;165:107337. doi: 10.1016/j.envint.2022.107337. Epub 2022 Jun 7. PMID 35696845
- [Result] Reiter EB, Escher BI, Rojo-Nieto E, Nolte H, Siebert U, Jahnke A. Characterizing the marine mammal exposome by iceberg modeling, linking chemical analysis and in vitro bioassays. Environ Sci Process Impacts. 2023 Nov 15;25(11):1802-1816. doi: 10.1039/d3em00033h. PMID 37132588
- See also: project website — http://www.ufz.de/exposo-meter